CLINICAL TRIAL: NCT01007201
Title: A Clinical Study to Assess the Immunogenicity and Safety of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in Healthy Subjects Aged Over 1 Year Old to 18 Years Old
Brief Title: Immunogenicity and Safety of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Jeffrey Chen / Vice President, Adimmune Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLU09002
Record Dates: First submitted 2009-11-01; First posted 2009-11-03 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: Influenza; H1N1; vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- H1N1 vaccine of 15 μg HA on Day 0 and 21 (Experimental): 15 μg HA (0.5 mL) per injection, 2 injections 50 children (aged over 3 years old to 6 years old) and 50 children/teenagers (aged over 6 years old to 18 years old) were assigned to receive two injections of H1N1 vaccine 3 weeks apart
  Interventions: Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated
- H1N1 vaccine of 7.5 μg HA on Day 0 and 21 (Experimental): 7.5 μg HA (0.25 mL) per injection, 2 injections 50 toddlers (aged over 1 year old to 3 years old) were assigned to receive two injections of H1N1 vaccine 3 weeks apart
  Interventions: Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated

INTERVENTIONS:
Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated
  Other Names: AdimFlu-S (A/H1N1)

SUMMARY:
This is a laboratory-blinded study in healthy toddlers, children, and teenagers designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 vaccine (AdimFlu-S). There are 3 age strata, and each contains at least 50 subjects: greater than or equal to 1 year to less than 3 years, greater than or equal to 3 years to less than 6 years, and greater than or equal to 6 years to less than 18 years. In each age strata, all eligible subjects received 2 injections of AdimFlu-S (A/H1N1) at a designated dosage level (7.5 μg, 15 μg and 15 μg for 1~<3, 3~<6 and 6~<18 years, respectively) at 3 weeks apart.

Following immunization, safety is measured by assessment of adverse events for 6 weeks following the first vaccination, serious adverse events and new-onset chronic medical conditions through 7 months post first vaccination, and reactogenicity to the vaccines for 7 days following each vaccination. Immunogenicity testing includes hemagglutination inhibition (HAI) testing on serum obtained before first vaccination, and three and six weeks after first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls aged ≧ 1 year old to 18 years old on the day of first vaccination;
* Subject and/or parents(s)/legal guardian(s) was willing to comply with planned study procedures and be available for all study visits;
* Subject was in good physical health on the basis of medical history, physical examination;
* Subject and/or parents(s)/legal guardian(s) must read and signed the study-specific informed consent prior to initiation of any study procedure.

Exclusion Criteria:

* Subject ever received influenza vaccine within the previous 6 months;
* History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication (AdimFlu-S (A/H1N1));
* Personal or family history of Guillain-Barré Syndrome;
* An acute febrile illness within the last 72 hours prior to vaccination;
* Subject with bleeding disorder or has any coagulation disorder that needs receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular injection;
* Subjects with influenza-like illness as defined by the presence of fever (temperature ≧38.5℃ ) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
* Female subjects who are pregnant, lactating or likely to become pregnant during the study; Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study;
* Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
* Immunodeficiency, immunosuppressive or household contact with immunosuppression;
* History of wheezing or bronchodilator use within 3 months prior to study vaccine;
* Receipt of live virus vaccine within 1 month prior to study vaccination or expected receipt within 2 months after first study vaccination;
* Receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected receipt vaccination within 3 weeks after the immunogenicity evaluation period;
* Receipt of any blood products, including immunoglobulin in the prior 3 months;
* Underlying condition in the investigator's opinion may be inappropriate for vaccination;
* Significant chronic illness for which inactivated influenza vaccine is recommended or commonly used.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary immunogenicity objective is to assess the antibody response following a single dose of study vaccine, grouped by age of recipient, when administered at the 7.5 or 15 μg HA doses.
The primary safety objective of this study is to assess the safety of the study vaccine when administered at the 7.5 or 15 μg HA doses.

SECONDARY OUTCOMES:
The secondary immunogenicity objective is to assess the antibody response following 2 doses of study vaccine, grouped by age of recipient, when administered at the 7.5 or 15 μg HA doses.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ming Huang, Principal Investigator — National Taiwan University Hospital; Tzou-Yien Lin, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan Hsien